CLINICAL TRIAL: NCT02455557
Title: A Phase II Study of the Safety and Efficacy of SVN53-67/M57-KLH (SurVaxM) in Survivin-Positive Newly Diagnosed Glioblastoma
Brief Title: SurVaxM Vaccine Therapy and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 259614; NCI-2015-00694 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 259614 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2015-05-22; First posted 2015-05-28 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — montanide ISA 51; sargramostim; Colony-Stimulating Factors; Temozolomide

ARMS (1):
- Treatment (SurVaxM, temozolomide) (Experimental): Patients receive the first priming dose of SVN53-67/M57-KLH peptide vaccine in emulsion with montanide ISA 51 SC and sargramostim SC within 7-28 days after completion of chemoradiation. Treatment repeats every 2 weeks for a total of 4 doses in the vaccine priming phase and then every 12 weeks during the adjuvant phase in the absence of disease progression or unacceptable toxicity. Patients also receive standard adjuvant temozolomide PO or IV on days 1-5. Treatment repeats every 28 days for 6 courses or more (at the discretion of the investigator) in the absence of disease progression or unacceptable toxicity. Patients may then receive maintenance SVN53-67/M57-KLH peptide vaccine in emulsion with montanide ISA 51 SC and sargramostim SC every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Montanide ISA 51 VG; Biological: Sargramostim; Biological: SVN53-67/M57-KLH Peptide Vaccine; Drug: Temozolomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Montanide ISA 51 VG — Given SC
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: SVN53-67/M57-KLH Peptide Vaccine — Given SC
Drug: Temozolomide — Given PO or IV
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase II trial studies the side effects and how well vaccine therapy works when given together with temozolomide in treating patients with newly diagnosed glioblastoma. Vaccines made from the survivin peptide or antigen may help the body build an effective immune response to kill tumor cells that express survivin. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether temozolomide is more effective with or without vaccine therapy in treating glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate 6-month progression-free survival (PFS6) in patients with survivin positive newly diagnosed glioblastoma multiforme (GBM) treated with at least 4 doses of SVN53-67/M57-keyhole limpet hemocyanin (KLH) peptide vaccine (SurVaxM) and standard of care temozolomide.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of SurVaxM in patients receiving standard care adjuvant temozolomide.

II. To evaluate overall survival (OS) in patients with survivin positive newly diagnosed GBM treated with SurVaxM and adjuvant temozolomide.

III. To describe the immune response in patients treated with SurVaxM and predictors of response.

IV. To evaluate objective tumor response rate (applicable only for patients with evaluable disease at study entry, as defined per Response Assessment in Neuro-Oncology [RANO] criteria) and predictors of response.

OUTLINE:

Patients receive the first priming dose of SVN53-67/M57-KLH peptide vaccine in emulsion with montanide ISA 51 subcutaneously (SC) and sargramostim SC within 7-28 days after completion of chemoradiation. Treatment repeats every 2 weeks for a total of 4 doses in the vaccine priming phase and then every 12 weeks during the adjuvant phase in the absence of disease progression or unacceptable toxicity. Patients also receive standard adjuvant temozolomide orally (PO) or intravenously (IV) on days 1-5. Treatment repeats every 28 days for 6 courses or more (at the discretion of the investigator) in the absence of disease progression or unacceptable toxicity. Patients may then receive maintenance SVN53-67/M57-KLH peptide vaccine in emulsion with montanide ISA 51 SC and sargramostim SC every 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a Karnofsky performance status >= 70 (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Documented survivin-positive tumor status
* Pathologically confirmed diagnosis of glioblastoma multiforme (GBM); or World Health Organization (WHO) grade IV [gliosarcoma]
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hgb) > 9.0 g/dL
* Serum total bilirubin: =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 4.0 x ULN
* Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight [LMW] heparin) must meet the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Creatinine =< 1.8 mg/dl
* Human leukocyte antigen (HLA)-A*02, HLA-A*03, HLA-A*11 or HLA-A*24 positive patients
* No evidence of progressive disease from the postoperative period to the post-chemoradiation period, based on changes in the neurologic exam, steroid use, or evident radiographic progression, according to RANO criteria; Patients with increased or new gadolinium enhancement may continue on protocol if in the investigator's judgment that enhancement is likely due to pseuodoprogresion. The use of correlative imaging studies (including PWI) or diffusion weighted imaging (DWI) and repeat imaging after an interval of 2-4 weeks is strongly encouraged to help distinguish between pseudoprogression and true progression.
* Magnetic resonance imaging (MRI) (ideally completed within 96 hours after surgery) documenting gross total resection consisting of no gadolinium enhancement; or subtotal resection consisting of linear enhancement with (or without) nodular gadolinium enhancement measuring no greater than 1 cm x 1 cm x 1 cm total volume or 100 mm^2 in cross sectional area
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry, and have a negative pregnancy test prior to starting study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Dexamethasone dose less than or equal to 4 mg daily at time of study enrollment
* Patients must have completed initial radiation therapy (RT) and temozolomide (TMZ) for the treatment of their glioblastoma (i.e., completed 6-week course of RT and, completed >= 75% of 6-week course of induction TMZ chemotherapy)
* Participant must understand the investigational nature of this study and sign an independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* The patient must not have received any immunotherapy for their brain tumor
* Patients with serious concurrent infection or medical illness, which in the treating physician's opinion would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
* Patients who are pregnant or breast-feeding
* Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents) other than temozolomide
* Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin; patients who have been free of disease (any prior malignancy) for at least 3 years are eligible for this study
* Patients who have had repeat craniotomy for tumor therapy after receiving RT and TMZ treatment
* Patients who received other chemotherapeutics or investigational agents in addition to their radiation therapy and concomitant temozolomide treatment
* Patients who have received Gliadel wafers or alternating electrical field therapy (ETTF) are not eligible for this study
* Known history of an autoimmune disorder
* Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness
* Patients who have contraindication to MRI
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2025-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fenstermaker, Principal Investigator — Roswell Park Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Ahluwalia MS, Reardon DA, Abad AP, Curry WT, Wong ET, Figel SA, Mechtler LL, Peereboom DM, Hutson AD, Withers HG, Liu S, Belal AN, Qiu J, Mogensen KM, Dharma SS, Dhawan A, Birkemeier MT, Casucci DM, Ciesielski MJ, Fenstermaker RA. Phase IIa Study of SurVaxM Plus Adjuvant Temozolomide for Newly Diagnosed Glioblastoma. J Clin Oncol. 2023 Mar 1;41(7):1453-1465. doi: 10.1200/JCO.22.00996. Epub 2022 Dec 15. PMID 36521103

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (SurVaxM, Temozolomide)
Started | 66
Completed | 64
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (SurVaxM, Temozolomide)
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 61
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The 6-month progression-free survival (PFS6) estimated using the Kaplan-Meier methods. PFS6 is defined as the percentage of patients without tumor progression or death from any cause 6 months after the date of diagnosis by biopsy. Corresponding confidence intervals will be computed.
Time Frame: Date of diagnosis to the date of first observed disease progression or death due to any cause, assessed at 6 months
Population: All treated and eligible patients that completed the priming dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SurVaxM, Temozolomide)
Number analyzed (Participants) | 64
percentage of participants | 95 [86 to 98]

2. Secondary Outcome: Immune Responses to SurVaxM and Predictors of Response
Description: A series of exploratory analyses will initially take place including individual subject-level profile plots and overall mean plots used to examining the mean structure. Formal statistical examination of longitudinal patterns will be done through the use of a mixed model. Restricted maximum likelihood estimation will be utilized in the model fitting procedures. Once the model is fit, specific linear contrasts based on the estimated model parameters will be constructed and used to test hypotheses concerning between time point comparisons.
Time Frame: Up to 30 days after completion of study treatment
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Grade 3 or 4 Toxicities, According to National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4
Description: Toxicities will be summarized using simple frequencies by grade. CTEP Version 4 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) will be utilized for AE reporting. Results are presented for the number of participants with drug-related Grade 3 or 4 toxicity/adverse event (AE). Grades range from 0 (none) to 5 (death), with Grade 3 and 4 being defined as follows:
  Grade 0 = No AE; Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
Time Frame: Up to 30 days after completion of study treatment
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SurVaxM, Temozolomide)
Number analyzed (Participants) | 66
Participants
  Grade 1 | 13
  Grade 2 | 20
  Grade 3 | 29
  Grade 4 | 3
  Grade 5 | 1

4. Secondary Outcome: Overall Survival
Description: The median overall survival estimated using the Kaplan-Meier methods. Estimates of quantities such as median survival will be obtained. Corresponding confidence intervals will be computed.
Time Frame: Date of diagnosis until (1) date of death or (2) the last date patient known alive (if death is not observed), assessed up to 2 years
Population: All treated and eligible patients that completed priming dose
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (SurVaxM, Temozolomide)
Number analyzed (Participants) | 64
months | 25.8 [19.5 to 43.5]

ADVERSE EVENTS:
Time Frame: Start date of intervention until 30 days after the last intervention or until the event has resolved, the study participant is lost to follow-up, the start of a new treatment, or until the study investigator assesses the event(s) as stable or irreversible, will be reported.
Arm/Group | Treatment (SurVaxM, Temozolomide)
All-Cause Mortality (participants affected / at risk) | 36/66
Serious Adverse Events (participants affected / at risk) | 22/66
Other Adverse Events (participants affected / at risk) | 65/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SurVaxM, Temozolomide) (N=66)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 3 (4)
Confusional state (Psychiatric disorders) | 5 (6)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Chest tube insertion (Surgical and medical procedures) | 1 (1)
Craniotomy (Surgical and medical procedures) | 2 (2)
Hip surgery (Surgical and medical procedures) | 1 (1)
Thoracotomy (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SurVaxM, Temozolomide) (N=66)
Anaemia (Blood and lymphatic system disorders) | 12 (41)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (7)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (9)
Deafness (Ear and labyrinth disorders) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4)
Cushingoid (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 18 (20)
Diarrhoea (Gastrointestinal disorders) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 31 (48)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (21)
Application site discolouration (General disorders) | 1 (1)
Asthenia (General disorders) | 5 (5)
Chills (General disorders) | 2 (3)
Cyst (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 30 (45)
Gait disturbance (General disorders) | 4 (4)
Implant site oedema (General disorders) | 1 (1)
Influenza like illness (General disorders) | 3 (8)
Injection site bruising (General disorders) | 4 (5)
Injection site discharge (General disorders) | 1 (1)
Injection site erythema (General disorders) | 2 (2)
Injection site induration (General disorders) | 3 (6)
Injection site inflammation (General disorders) | 1 (1)
Injection site nodule (General disorders) | 1 (1)
Injection site pain (General disorders) | 9 (14)
Injection site pruritus (General disorders) | 4 (5)
Injection site rash (General disorders) | 1 (1)
Injection site reaction (General disorders) | 27 (65)
Injection site swelling (General disorders) | 3 (3)
Malaise (General disorders) | 2 (4)
Mucosal inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 6 (10)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Injection site infection (Infections and infestations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (8)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (7)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (3)
Alanine aminotransferase increased (Investigations) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (4)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2)
Blood glucose increased (Investigations) | 1 (1)
Blood ketone body (Investigations) | 1 (1)
Haemoglobin urine present (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 21 (92)
Neutrophil count decreased (Investigations) | 15 (55)
Neutrophil count increased (Investigations) | 4 (10)
Platelet count decreased (Investigations) | 25 (66)
Transaminases increased (Investigations) | 1 (1)
Urine ketone body present (Investigations) | 1 (1)
Weight decreased (Investigations) | 3 (3)
Weight increased (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 21 (103)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 18 (22)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (8)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amnesia (Nervous system disorders) | 2 (2)
Aphasia (Nervous system disorders) | 5 (6)
Ataxia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 4 (4)
Coordination abnormal (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (14)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 20 (25)
Hemiparesis (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2)
Mental impairment (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 5 (6)
Partial seizures (Nervous system disorders) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 11 (12)
Seizure like phenomena (Nervous system disorders) | 2 (2)
Sinus headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (2)
Affect lability (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Confusional state (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 3 (4)
Dysphoria (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Libido decreased (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Incontinence (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 8 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 5 (5)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (5)
Rotator cuff repair (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 4 (6)
Hypotension (Vascular disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT02455557/Prot_SAP_000.pdf